CLINICAL TRIAL: NCT05739227
Title: Early Clinical Study of Allogenic CD19-CAR-NK Cells (JD001) in the Treatment of Refractory or Relapsed(r/r) B-cell Hematologic Malignancies
Brief Title: Safety and Efficacy of Allogenic CD19-CAR-NK Cells in Treatmenting r/r B-cell Hematologic Malignancies
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Kai Lin Xu，MD, Principal Investigator, Xuzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2022-KL252-01
Record Dates: First submitted 2023-02-11; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Acute Lymphoblastic Leukemia; B-cell Lymphoma; Chronic Lymphocytic Leukemia
Keywords: B-cell hematologic malignancies; allogenic CD19-CAR-NK cells
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- allogenic CD19-CAR-NK (Experimental): Enrolled patients will receive prespecified dose of allogenic CD19-CAR-NK cells.
  Interventions: Other: allogenic CD19-CAR-NK cells

INTERVENTIONS:
Other: allogenic CD19-CAR-NK cells — The relapsed/refractory B-cell hematologic malignancies patients will receive allogenic CD19-Targeted CAR-NK cells infusion up to 3 dose levels (1x10^6/kg, 5x10^6/kg, 2x10^7/kg) after FCE chemotherapy

SUMMARY:
This is an open label, single-arm, Phase I study to evaluate the efficacy and safety of allogenic CD19-CAR-NK cells in subjects with refractory or relapsed B-cell hematologic malignancies. A leukapheresis procedure will be performed to manufacture Anti-CD19 chimeric antigen receptor (CAR) modified NK cells. Prior to allogenic CD19-CAR-NK cells infusion subjects will receive lymphodepleting therapy with fludarabine, cyclophosphamide and etoposide.

DETAILED DESCRIPTION:
This open label, single-arm, Phase I study aims to evaluate the efficacy and safety of allogenic CD19-CAR-NK cells in subjects with refractory or relapsed B-cell hematologic malignancies. A leukapheresis procedure will be performed to manufacture Anti-CD19 chimeric antigen receptor (CAR) modified NK cells. Prior to allogenic CD19-CAR-NK cells infusion subjects will receive lymphodepleting therapy with fludarabine, cyclophosphamide and etoposide. After infusion, the investigators will observe the characteristics of dose limited toxicity (DLT), and determine the maximum tolerable agent MTD and rp2d were confirmed. To provide basis for the dosage and treatment plan of cell products in follow-up clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Age18-75years old, no gender or race;
2. Expected survival period ≥ 3 months;
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2;
4. Confirmed relapsed/refractory B-cell tumor and tumor cells expressing CD19, including acute B-cell lymphoblastic leukemia and B-cell lymphoma; and meets the following criteria for refractory or relapsed B-cell hematologic malignancies: (1) Refractory or relapsed acute B-cell lymphoblastic leukaemia (meets one of the following four criterias): a.Relapse within 6 months after the initial remission; b. Initial refractory patients with failure to achieve complete remission(CR) after 2 cycles of standard chemotherapy; c.Failure to achieve CR or relapse after first line or multiline salvage chemotherapy; d.Patients who are not fitable for hematopoietic stem cell transplantation (HCT), or give up HCT due to limitations, or relapse after HCT.(2) Refractory or relapsed B-cell lymphoma (meets 1 of the following first 4 criterias plus the fifth): a.≤50% decrease in SPD of up to 6 target measurable nodes and extranodal sites or disease progression after 4 cycles of standard chemotherapy; b.Relapse within 6 months after CR; c.Two or more times relapse after CR; d.Subjects who are not fitable for HCT, or give up HCT due to limitations, or relapse after HCT; e.Subjects must be treated with adequate treatment, including at least monoclonal antibodies against CD20 or combination chemotherapy containing anthracyclines;
5. Measurable lesions meets at least one of the following requirements during screening: (1) For lymphoma patients, the length of a single lesion ≥15mm or two or more lesions with the length ≥10mm; (2) Acute B-cell lymphoblastic leukaemia patients with persistent positive MRD or relapse with positive MRD;
6. Within 3 days prior to initial treatment, the organ functions meet the following requirements: (1) complete blood cell count: a.Absolute neutrophil counts ≥ 1.0 ×10^9/L and not treated with G-CSF within 7 days; b.Hemoglobin ≥6g/dL(red blood cell transfusion is permitted); c.Platelet ≥50×10^9/L, (platelet transfusion is permitted);(2) Liver function: alanine transaminase (ALT)/ aspartate aminotransferase(AST) ≤ 3× times upper normal limit(ULN), total bilirubin ≤ 2 times ULN (direct bilirubin ≥1.5 times ULN is acceptable for subjects with Gilbert-Meulengracht syndrome);(3) Coagulation function: International standardized ratio (INR) or activated partial thrombin time (APTT) ≤1.5 times ULN; (4) Renal function: serum creatinine≤1.5×ULN or creatinine clearance rate ≥30mL/min; (5) Corrected serum calcium ≤14mg/dL (≤3.5mmol/L) or free calcium ≥6.5mg/dL(≥1.6mmol/L); (6) Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 50%;
7. Informed Consent/Assent: All subjects must have the ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

1. Central nervous system involved;
2. ≥2 grade persistent nonhematologic toxicity of associated with prior treatment;
3. Systemic steroid therapy exceeding the equivalent of ≥30mg/kg/day of prednisone within 48 hours prior to the first dose of study drug or other immunosuppressive therapies(except for topical and inhaled glucocorticoid therapy, or short-term prophylactic therapy with glucocorticoid);
4. Severe cardiovascular and cerebrovascular diseases, including: (1) Some cardiovascular and cerebrovascular diseases (such as congestive heart failure, acute myocardial infarction, unstable angina pectoris, stroke, transient ischemic attack, deep vein thrombosis or pulmonary embolism, etc.) occurr within 6 months prior to the first dose of study drug; (2)New York Heart Association (NYHA) Class ≥3 or uncontrolled malignant arrhythmias; (3)The researchers assessed that the subjects with other cardiovascular and cerebrovascular diseases are not suitable for the study;
5. Any active infection requiring systemic therapy by intravenous infusion within 14 days prior to the first dose of study drug, including: HBV, HCV, HIV, syphilis infection, or active pulmonary tuberculosis;
6. History of hypersensitivity reactions to murine protein-containing products, or macromolecular biopharmaceuticals such as antibodies or cytokines;
7. Previous or next organ transplant(except for HCT);
8. Women who are pregnant (urine/blood pregnancy test positive) or lactating;
9. Patients cannot guarantee effective contraception (condom or contraceptives, etc.) within 6 months after enrollment;
10. Any unstable condition potentially imperiling patient safety and compliance;
11. Known alcohol dependence or drug dependence;
12. According to the investigator's judgment, the patient has other unsuitable grouping conditions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities | 1 month
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Objective Response Rate(ORR) | 3 months
  Assessment of ORR (ORR = CR + CRi + PR) at 3 months of treatment

SECONDARY OUTCOMES:
Progression free survival(PFS) | Month 6,12
  Assessment of PFS at month 6,12
Overall Survival(OS) | Month 6, 12, 18 and 24
  Assessment of OS at month 6, 12, 18 and 24
Minimal-residual disease negative overall response rate(MRD-ORR) | Month 6, 12
  Assessment of MRD- ORR at month 6,12

CONTACTS AND LOCATIONS:
Overall Officials: Kailin Xu, M.D., Ph.D., Principal Investigator — Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China